CLINICAL TRIAL: NCT06118242
Title: The Effect of Chlorhexidine Gluconate, Sodium Bicarbonate, Ozonated Water and Hypochlorous Acid Solutions Used in Oral Care on Preventing Ventilator-Associated Pneumonia.
Brief Title: The Effect of Solutions Used in Oral Care on Preventing Ventilator-Associated Pneumonia.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Sercan Özdemir, Register Nurse, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AdnanMU-NDH-OZDEMIR-001
Record Dates: First submitted 2023-10-30; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Ventilator-Associated Pneumonia
Keywords: Oral Hygiene; Mechanical Ventilation; Intensive Care Units
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Results Related to Ventilator-Associated Pneumonia in Patients (Experimental): Use of 0.12% Chlorhexidine Gluconate,1% Chlorhexidine Gluconate, Sodium Bicarbonate, Ozonated Water and Hypochlorous Acid.
  Interventions: Other: Use of oral care solutions
- Results Regarding the Oral Mucous Membrane Integrity of Patients (Experimental): Use of 1% Chlorhexidine Gluconate, Sodium Bicarbonate, Ozonated Water and Hypochlorous Acid.
  Interventions: Other: Use of oral care solutions

INTERVENTIONS:
Other: Use of oral care solutions — Oral care solutions to be used: Chlorhexidine Gluconate, Sodium Bicarbonate, Ozonated Water and Hypochlorous Acid

SUMMARY:
The goal of this clinical trial is to learn about effects of chlorhexidine gluconate, sodium bicarbonate, ozonated water and hypochlorous acid solutions used in oral care of patients on mechanical ventilation support on preventing ventilator associated pneumonia.

The main question[s] it aims to answer are:

Is there any difference between 1% chlorhexidine gluconate, sodium bicarbonate, ozonated water and hypochlorous acid solutions versus 0.12% chlorhexidine gluconate solution used in oral care in preventing the development of VAP? Is there any difference between 1% chlorhexidine gluconate, sodium bicarbonate, ozonated water and hypochlorous acid solutions versus 0.12% chlorhexidine gluconate solution used in oral care in preventing the development of VAP?

Researchers will compare 1% chlorhexidine gluconate, sodium bicarbonate, ozonated water and hypochlorous acid solutions to see if VAP

DETAILED DESCRIPTION:
Many problems may develop in patients on mechanical ventilation support in intensive care units. The most important of these is ventilator-associated pneumonia (VAP) caused by inadequate oral care in patients on mechanical ventilator support. The aim of the thesis is to examine the effect of chlorhexidine gluconate, sodium bicarbonate, ozonated water and hypochlorous acid solutions used in oral care in preventing ventilator-associated pneumonia in patients on mechanical ventilation support.

This research was planned as a randomized controlled experimental study. The sample of the study will consist of 105 intubated adult patients hospitalized in the Anesthesia and Reanimation Intensive Care Unit of the Republic of Turkey Ministry of Health Aydın Provincial Health Directorate Nazilli State Hospital. Patients will be divided into a total of 5 groups: 4 experimental and 1 control group. The groups to which 1% chlorhexidine gluconate, sodium bicarbonate, ozonated water and hypochlorous acid solutions are applied will constitute the experimental group, and the patients who receive oral care with 0.12% chlorhexidine gluconate, which is routinely applied in the clinic, will constitute the control group. Patients will be given oral care by the nurse with determined solutions (chlorhexidine gluconate, sodium bicarbonate, ozonated water and hypochlorous acid) 4 times a day according to the oral care protocol, and the oral mucosa of all patient groups will be evaluated every morning for 7 days. A deep tracheal aspirate sample will be taken and a chest x-ray will be taken on the first and seventh days after hospitalization of intubated patients. The development of VAP in patients will be evaluated with the clinical pulmonary infection score.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age
* Being under mechanical ventilation treatment for at least 24 hours
* Agreeing to participate in the research

Exclusion Criteria:

* Patients who are extubated
* Patients transferred to another clinic
* Those who did not agree to participate in the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2023-11-15 (Estimated); Primary Completion 2024-11-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Ventilator associated pneumonia | one week
  We will used the commonly used clinical pulmonary infection score (CPIS), which includes temperature, leucocyte count and morphology, amount of tracheal secretions and their character, alveolar oxygen pressure (PaO2)/fraction of inspired oxygen (FiO2) ratio, findings of pulmonary infiltration and progression on chest X-ray, and growth of any pathogenic bacterial growth from the tracheal aspirate. Whereas the CPIS score of >6 or 6 suggests VAP.

CONTACTS AND LOCATIONS:
Overall Officials: Gülengün TÜRK, Prf. Dr, Study Director — Aydin Adnan Menderes University
Locations (1):
- Nazilli State Hospital, Aydin, Yesil, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No